CLINICAL TRIAL: NCT03882398
Title: Effects of a High-intensity Progressive-cycle Program on Quality of Life and Motor Symptomatology in Parkinson's Disease Population: a Pilot Randomized Controlled Trial
Brief Title: Effects of a High-intensity Progressive-cycle Program on Quality of Life and Motor Symptomatology in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vigo (Other)
Responsible Party: Principal Investigator, José M. Cancela, Principal Investigator, University of Vigo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2018
Record Dates: First submitted 2019-03-11; First posted 2019-03-20 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Parkinson Disease; Exercise; Physical Activity; Quality of Life
Keywords: Neurodegenerative disorders; physical activity; balance; endurance
MeSH Terms: conditions — Parkinson Disease; Motor Activity; Neurodegenerative Diseases

STUDY DESIGN:
Intervention Model Description: A pilot randomized controlled trial.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Fourteen patients were randomly assigned to the two groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The experimental group (EG) participated in a once a week physical exercise program for 8 weeks. The session consisted of balance training, followed by aerobic endurance training with exercise peddlers. At the beginning of the program, each session lasted 25 minutes and progressed to 35 minutes, in the last two weeks
  Interventions: Other: Balance; Other: Endurance
- Control Group (Active Comparator): The control group (CG) only performed routine balance exercises once a week (10 min)
  Interventions: Other: Balance

INTERVENTIONS:
Other: Balance — Balance program (10 minutes)
  Balance on bosu ball and ball drills Coordination in rings with single leg stance and ball drills Straight line walk with head up Straight line walk and hip flexion, knee flexion and head up
  (Duration: 10 minutes. Sets: 2 minutes per exercise. Rest: 30 seconds between exercises)
Other: Endurance — Progressive-cycle program (15-25 minutes)
  Warming up Pedalling with 0 resistance (2 minutes)
  Main Part* Week 1-2 : 3x2 minutes Week 3-4 : 4x2 minutes Week 5-6 : 5x2 minutes Week 7-8 : 6x2 minutes
  Return to resting stage Pedalling with 0 resistance (1 minute)
  (*Pedalling with resistance set at 3-4. Rest: 2 minutes between sets or 120 beats/minute. One more set added every two weeks and workout intensity maintained at 70% of heart rate reserve-HRR)
  Arms: Experimental group

SUMMARY:
TITLE: Effects of a high-intensity progressive-cycle program on quality of life and motor symptomatology in Parkinson's disease population

BACKGROUND: The benefits of aerobic exercise in persons with Parkinson's disease (PD) have been widely studied; however, little research has been done on the effect of high-intensity aerobic exercise in this group.

HYPOTHESIS: The high-intensity aerobic training in pedaliers, combined with balance training, improves motor symptoms and quality of life in a population with Parkinson Disease, Hoehn & Yahr 1-3.

OBJETIVES: To ascertain whether high-intensity aerobic training with exercise peddlers and balance training can improve motor symptoms and quality of life in a PD population of Hoehn &Yahr (H&Y) disability score 1-3.

METHODOLOGY Setting: Rehabilitation centers in secondary care. Design: A pilot randomized controlled trial. Participants: A total of 14 patients participated in the 8-week study. Interventions: They were comprised of a control group (n=7) that followed a balance protocol and an experimental group (n=7) that performed high intensity (70%) aerobic workout using an exercise peddler + a balance protocol once a week.

Main Outcome Measures: The primary outcome measures included the 8-Foot Up and Go, test, 6-minute walk test, test 2-minute step tets, Parkinson Disease Questionnaire-39 (PDQ39), Unified Parkinson's Disease Rating Scale (MDS-UPDRS) and Tinetti test.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Parkinson Disease, Hoehn & Yahr score of 1-3.

Exclusion Criteria:

* History or evidence of dementia or other neurological impairment/cardiovascular diseases that may affect the high-intensity endurance workout

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Sintomatology of Parkinson Disease | 12 weeks
  The Movement Disorders Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) evaluates the degree of symptomatology of the person with Parkinson's Disease. The total score range ranges from 0 to 200, with higher values indicating a greater impact of the symptoms. Each item is scored from 0 to 4, with 0 being the least and 4 the most severe. The scores are added.
Quality of life in Parkinson Disease: PDQ39 | 12 weeks
  The quality of life questionnaire for Parkinson's disease is a specific questionnaire that evaluates the quality of life, where a lower score means that the patient has a better quality of life. It consists of 39 questions, and its value is expressed in percentages, the percentages closest to zero express a better quality of life. In addition, their results can also be expressed in 8 different areas (mobility, activities of daily life, stigma, emotional well-being, social support, communication, body discomfort, cognitive impairment), which are interpreted in the same way.
Physical Conditions | 12 weeks
  The Senior Fitness Test, is a battery of 7 tests to evaluate the physical state of the elderly, and has been validated for people with Parkinson's Disease. This battery evaluates the strength of lower and upper limbs with the 30 seconds chair stand and arm curl tests, to more repetitions, more strength. It also evaluates the flexibility of both lower and upper limbs with the chair sit and reach and back stractch tests, which are measured in centimeters, to more centimeters greater flexibility. Aerobic endurance is assessed by means of the 6 minute walk test that is measured in meters, and the 2 minute step test that is measured in cycles. The more number of cycles and meters, the better aerobic resistance. The balance is evaluated by means of the 8 foot up and go test, which is measured in seconds, and the less the better the balance. These results by means of a mathematical formula give an absolute value that to higher score better physical condition
Balance | 12 weeks
  Tinetti test The objective of the Tinetti test is to evaluate the possible alterations of balance in a population of elderly people. The test consists of two parts: nine elements of balance and six elements of march. The maximum total score is 28, and would mean that gait and balance are normal

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Vigo, Pontevedra, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886